CLINICAL TRIAL: NCT04241068
Title: Phase 3b Open-Label, Multicenter, Safety Study of BIIB037 (Aducanumab) in Subjects With Alzheimer's Disease Who Had Previously Participated in the Aducanumab Studies 221AD103, 221AD301, 221AD302 and 221AD205
Brief Title: A Study to Evaluate Safety and Tolerability of Aducanumab in Participants With Alzheimer's Disease Who Had Previously Participated in the Aducanumab Studies 221AD103, 221AD301, 221AD302 and 221AD205
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 221AD304; 2019-004368-22 (EudraCT Number)
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aducanumab (Experimental): Participants will be administered aducanumab 10 milligrams per kilogram (mg/kg) by intravenous (IV) infusions every four weeks (Q4W) for a duration of 100 weeks during the Core Treatment Period. Eligible participants will continue to receive aducanumab 10 mg/kg IV infusion, Q4W, for 52 weeks during the Long-Term Extension (LTE) Treatment Period.
  Interventions: Drug: Aducanumab

INTERVENTIONS:
Drug: Aducanumab — Administered as specified in the treatment arm.
  Other Names: BIIB037

SUMMARY:
The primary objective is to evaluate the safety and tolerability of aducanumab over 100 weeks of treatment after a wash-out period imposed by discontinuation of feeder studies in participants who had previously received aducanumab (i.e. previously treated participants) or who had previously received placebo (i.e. treatment-naïve participants).

ELIGIBILITY:
Key Inclusion Criteria:

Core Treatment Period:

* Participant was participating in an aducanumab clinical study at the time of the announcement of early termination (feeder studies).
* Has one care partner who, in the Investigator's opinion, has adequate contact with the participant as to be able to provide accurate information about the participant's cognitive and functional abilities.

LTE Treatment Period:

* Participant must have completed the Core study period (Week 102) and adequately tolerated 10 mg/kg of aducanumab during the Core study period in the opinion of the Investigator.
* Has one informant/care partner who, in the Investigator's opinion, has frequent and sufficient contact with the participant as to be able to provide accurate information about the participant's cognitive and functional abilities.

Key Exclusion Criteria:

Core Treatment Period:

* Any medical or neurological condition (other than Alzheimer's Disease) that might be a contributing cause of the participant's cognitive impairment.
* Stroke or any unexplained loss of consciousness within 1 year prior to Screening.
* Clinically significant unstable psychiatric illness in past 6 months.
* History of unstable angina, myocardial infarction, advanced chronic heart failure, or clinically significant conduction abnormalities within 1 year prior to Screening.
* A seizure event that occurred after the last visit of the feeder study and before Screening for this study.
* Evidence of impaired liver function as shown by an abnormal liver function profile at Screening.
* History of or known seropositivity for HIV.
* Clinically significant systemic illness or serious infection within 30 days prior to or during Screening.
* Contraindications to having a brain magnetic resonance imaging (MRI).

LTE Treatment Period:

* Any medical or psychiatric contraindication or clinically significant abnormality that, in the opinion of the Investigator, will substantially increase the risk associated with the participant's enrollment in and completion of the study.

Note- Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1696 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (293):
- United States (103):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Dignity Health, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - UCI MIND, Irvine, California
  - University of California San Diego Medical Center, La Jolla, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - USC Keck School of Medicine, Los Angeles, California
  - Mary S. Easton Center for Alzheimer's Disease Research, UCLA, Los Angeles, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Anderson Clinical Research, Redlands, California
  - Pacific Research Network, Inc, San Diego, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research Medical Group Inc., Sherman Oaks, California
  - University of Colorado Denver, Aurora, Colorado
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Yale University, Fairfield, Connecticut
  - Invicro, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Georgetown University Clinical Research Unit (CRU), Washington D.C., District of Columbia
  - JEM Research, Atlantis, Florida
  - Bradenton Research Center, Inc, Bradenton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami Jewish Health System, Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Accelerated Enrollment Solutions (AES), Orlando, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Quantum Laboratories Inc., Pompano Beach, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Emory University Cognitive Neurology Clinic & ADRC, Atlanta, Georgia
  - Medical Research Health and Education Foundation, Inc, Columbus, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Alexian Brothers Medical Center - Neuroscience Research Institute, Elk Grove Village, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson, Wallack, Munshower Neurology, P.C., Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Fairway, Kansas
  - Ascension Via Christi Research, a division of Ascension Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - McLean Hospital, Belmont, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital Department of Neurology, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Mayo Clinic, Rochester, Michigan
  - Hattiesburg Clinic, PA, Hattiesburg, Mississippi
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Advanced Memory Research Inst. of NJ, PC, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Empire Neurology, PC, Latham, New York
  - New York University Medical Center PRIME, New York, New York
  - Weill Cornell Medical College (WCMC) - Judith Jaffe Multiple Sclerosis Center (JJMSC), New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - AMC Research, LLC, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Gastroenterology Associates of the Piedmont, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Northeastern Pennsylvania Memory and Alzheimer's Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - Senior Adult Specialty Research, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - University of Washington Medical Centre, Seattle, Washington
  - Kingfisher Cooperative, LLC, Spokane, Washington
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Australia (8):
  - The Prince Charles Hospital, Chermside, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research (Erina), Erina, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg West, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Austria (3):
  - LKH - Universitaetsklinikum Graz, Graz
  - Christian-Doppler-Klinik - Universitätsklinikum Salzburg, Salzburg
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (7):
  - AZ Klina, Brasschaat
  - AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Canada (17):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - The Medical Arts Health Research Group, Kamloops, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - UBC Hospital, Vancouver, British Columbia
  - Medical Arts Health Research Group, West Vancouver, British Columbia
  - True North Clinical Research - Halifax Inc., Halifax, Nova Scotia
  - True North Clinical Research, Kentville, Nova Scotia
  - St. Joseph's HC- Parkwood Institute, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - Institut et Clinique MoCA, Greenfield Park, Quebec
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Denmark (3):
  - CCBR - Ålborg - DK, Aalborg
  - Danish Dementia Research Centre, Copenhagen
  - CCBR - Vejle - DK, Vejle
- Finland (3):
  - Terveystalo Ruoholahti, Helsinki
  - Itä-Suomen yliopisto, Aivotutkimusyksikkö, Kuopio
  - CRST, Clinical Research Services Turku, Turku
- France (15):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hopital Purpan, Toulouse, Haute Garonne
  - Hôpital La Grave, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Nantes - Hopital Nord Laënnec, Nantes, Loire Atlantique
  - CHU Reims - Hôpital Maison Blanche, Reims, Marne
  - CHU Lille - Hopital Roger Salengro, Lille, Nord
  - Hôpital Lariboisière, Paris, Paris
  - CHU de Lyon - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - Hôpital des Chapennes, Villeurbanne, Rhone
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Broca, Paris
- Germany (22):
  - Studienzentrum fur Neurologie und Psychiatrie, Böblingen, Baden-Wurttemberg
  - ISPG - Institut fuer Studien zur Psychischen Gesundheit, Mannheim, Baden-Wurttemberg
  - mind mvz GmbH, Stuttgart, Baden-Wurttemberg
  - Neuropoint Studienzentrum, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH- Hohe Warte, Bayreuth, Bavaria
  - Bezirkskrankenhaus Guenzburg, Günzburg, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Institut fuer Schlaganfall- und Demenzforschung (ISD), München, Bavaria
  - Neuropraxis Muenchen Sued, Unterhaching, Bavaria
  - Neuro Centrum Science GmbH, Geschaftführende Gesellschafterin Barbara Unsorg und Prüfarzt Dr. med. G, Erbach im Odenwald, Hesse
  - Neurologische Gemeinschaftspraxis Kassel, Kassel, Hesse
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Universitaetsklinikum Aachen AOeR, Aachen, North Rhine-Westphalia
  - Neurozentrum Bielefeld, Bielefeld, North Rhine-Westphalia
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Zentrum f. Neurologisch- Psychiatrische Studien und Begutachtung, Siegen, North Rhine-Westphalia
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - Emovis GmbH, Berlin
  - Neurologie im Tempelhofer Hafen, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Berlin Buch, Berlin
- Italy (16):
  - Ospedale degli Infermi, Ponderano, Biella
  - Azienda Ospedaliera Card. G. Panico, Tricase, Lecce
  - ASST di Monza, Monza, Milano
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - AOU dell'Università degli studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera e Universitaria di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Fondazione Santa Lucia IRCCS, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (33):
  - Research Site, Obu-shi, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Inzai-shi, Chiba
  - Research Site, Toon-shi, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Aizu-Wakamatsu, Fukushima
  - Research Site, Otake-shi, Hiroshima
  - Research Site, Asahikawa-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Himeji-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kita-gun, Kagawa-ken
  - Research Site, Kamakura-shi, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Tsu, Mie-ken
  - Research Site, Togitsu, Nagasaki
  - Research Site, Nagaoka-shi, Niigata
  - Research Site, Yufu-shi, Oita Prefecture
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Tsukuba, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Iruma-gun, Saitama
  - Research Site, Kasukabe-shi, Saitama
  - Research Site, Shizuka-shi, Shizuoka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Bunkyō City, Tokyo-To
  - Research Site, Kiyose-shi, Tokyo-To
  - Research Site, Kodaira-shi, Tokyo-To
  - Research Site, Yamagata, Yamagata
- Netherlands (3):
  - Brain Research Center, Amsterdam
  - Amphia Ziekenhuis, Molengracht, Breda
  - Erasmus Medisch Centrum, Rotterdam
- Poland (12):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - PALLMED Sp. z o.o., Bydgoszcz
  - Klinika Psychiatrii Doroslych UCK, Gdansk
  - Novo-Med Zielinski i wspolnicy Sp. j., Katowice
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - NZOZ "NEURO-KARD", "Ilkowski i Partnerzy" Sp. Partn. Lek., Poznan
  - Neuro-Care Gabriela Klodowska, Siemianowice Śląskie
  - Centrum Medyczne Senior, Sopot
  - Osrodek Badan Klinicznych EUROMEDIS, Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra E.P.E - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital Beatriz Ângelo, Loures
  - CNS-Campus Neurologico Senior, Torres Vedras
- South Korea (6):
  - Inha University Hospital, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (14):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Policlinica Gipuzkoa, Donostia / San Sebastian, Guipuzcoa
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CAE Oroitu, Getxo, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Santa Maria, Lleida
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (4):
  - Skånes Universitetssjukhus, Malmo
  - Sahlgrenska Universitetssjukhuset, Mölndal Sjukhus, Mölndal
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (5):
  - Spitalzentrum Biel, Biel/Bienne
  - Hôpitaux Universitaires de Geneve- HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Regionale di Lugano, Lugano
  - Institut fur Regenerative Medizin-IREM Universitat Zurich, Campus Schlieren, Schlieren
- Taiwan (5):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (10):
  - Re:Cognition Health Ltd (London), London, Greater London
  - Charing Cross Hospital, London, Greater London
  - The National Hospital for Neurology and Neurosurgery Centre, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - The University of Edinburgh, Edinburgh, Lothian Region
  - The RICE Centre, Bath, Somerset
  - Queen Elizabeth University Hospital Campus, Glasgow, Strathclyde
  - Glasgow Memory Clinic Ltd, Motherwell, Strathclyde
  - Ninewells Hospital, Dundee, Tayside Region
  - Newcastle University, Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the investigative sites in the United States, Australia, Austria, Belgium, Canada, Denmark, Finland, France, Germany, Italy, Japan, South Korea, Netherlands, Poland, Portugal, Spain, Sweden, Switzerland, Taiwan, and United Kingdom from 02 Mar 2020 to 22 Jul 2024.
Pre-assignment Details: A total of 1696 participants were enrolled and treated in the core period, of which 1118 participants completed the core period. Out of the participants who completed the core period, 1041 participants entered the long-term extension (LTE) period, and 508 participants completed the LTE period.
Groups:
- Aducanumab: Participants were administered aducanumab 10 milligrams per kilogram (mg/kg) by intravenous (IV) infusions every four weeks (Q4W) for 100 weeks during the Core Treatment Period. Eligible participants continued to receive aducanumab 10 mg/kg IV infusion, Q4W, for 52 weeks during the LTE Treatment Period.
Period: Core Treatment Period
Arm/Group | Aducanumab
Started | 1696
Completed | 1118
Not Completed | 578
Not completed — Adverse Event | 91
Not completed — Change of Treatment | 4
Not completed — Consent Withdrawn | 143
Not completed — Death | 26
Not completed — Disease Progression | 67
Not completed — Investigator Decision | 40
Not completed — Loss of Capacity | 9
Not completed — Lost to Follow-up | 11
Not completed — Relocation | 4
Not completed — Study Terminated by Sponsor | 1
Not completed — Study Visit Burden | 40
Not completed — Withdrawal by Guardian/caretaker | 99
Not completed — Missing | 2
Not completed — Reason Not Specified | 41
Period: LTE Period
Arm/Group | Aducanumab
Started (77 participants were not eligible for LTE period.) | 1041
Completed | 508
Not Completed | 533
Not completed — Adverse Event | 19
Not completed — Change of Treatment | 1
Not completed — Consent Withdrawn | 71
Not completed — Death | 8
Not completed — Disease Progression | 11
Not completed — Investigator Decision | 12
Not completed — Loss of Capacity | 2
Not completed — Lost to Follow-up | 7
Not completed — Relocation | 6
Not completed — Site Terminated by Sponsor | 26
Not completed — Study Terminated by Sponsor | 276
Not completed — Study Visit Burden | 10
Not completed — Withdrawal by Guardian/caretaker | 19
Not completed — Reason Not Specified | 65

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) population included all participants who had received at least one dose of aducanumab in the study 221AD304.
Groups:
- Aducanumab: Participants were administered aducanumab 10 mg/kg by IV infusions, Q4W for 100 weeks during the Core Treatment Period. Eligible participants continued to receive aducanumab 10 mg/kg IV infusion, Q4W, for 52 weeks during the LTE Treatment Period.
Arm/Group | Aducanumab
Number analyzed (Participants) | 1696
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 881
  Male | 815
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 185
  Race: Black or African American | 8
  Race: White | 1399
  Race: Not Reported Due to Confidentiality Regulations | 55
  Race: Other | 3
  Race: Unknown | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 61
  Ethnicity: Not Hispanic or Latino | 1562
  Ethnicity: Not Reported Due to Confidentiality Regulations | 73

OUTCOME MEASURES:

1. Primary Outcome: Core Treatment Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a participant/clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal(investigational) product, whether or not related to medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in significant disability/incapacity or congenital anomaly, is medically important event. TEAE or Serious TEAEs are defined as any AE that has an onset date and time that is on or after date and time of first dose of study treatment, or that has worsened after date and time of first dose of study treatment.
Time Frame: From the first dose of study drug to end of follow-up (up to Week 118)
Population: The safety population for the core period included all participants who had received at least one dose of aducanumab in the core period.
Measure: Count of Participants; unit: Participants
Groups:
- Aducanumab: Participants were administered aducanumab 10 mg/kg by IV infusions, Q4W for 100 weeks during the Core Treatment Period.
Arm/Group | Aducanumab
Number analyzed (Participants) | 1696
Participants
  TEAEs | 1549
  Serious TEAEs | 318

2. Primary Outcome: Core Treatment Period: Number of Participants With AEs Leading to Treatment Discontinuation (TD) and Study Withdrawal (SW)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From the first dose of study drug to end of follow-up (up to Week 118)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aducanumab
Number analyzed (Participants) | 1696
Participants
  AEs leading to TD | 168
  AEs leading to SW | 129

3. Primary Outcome: Core Treatment Period: Number of Participants With Amyloid-Related Imaging Abnormality-Edema (ARIA-E)
Description: Number of participants diagnosed with ARIA edema are reported.
Time Frame: Up to Week 118
Population: The safety magnetic resonance imaging (MRI) population for the core period included all participants who had received at least one dose of aducanumab in the core period and had at least one post-baseline MRI assessment in the core period. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aducanumab
Number analyzed (Participants) | 1656
Participants | 422

4. Primary Outcome: Core Treatment Period: Number of Participants With Amyloid-Related Imaging Abnormality- Hemorrhage or Superficial Siderosis (ARIA-H)
Description: Number of participants diagnosed with ARIA hemmorrhage or superficial siderosis are reported.
Time Frame: Up to Week 118
Population: The safety MRI population for the core period included all participants who had received at least one dose of aducanumab in the core period and had at least one post-baseline MRI assessment in the core period. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aducanumab
Number analyzed (Participants) | 1656
Participants | 505

5. Primary Outcome: Core Treatment Period: Number of Participants With Positive Antidrug Antibodies (ADAs) in Serum
Description: The presence of serum ADAs was determined using a validated assay. A standard 3-tiered approach was used including screening assay, confirmatory assay, and titration assay. The number of participants with a positive response to ADAs are reported.
Time Frame: Up to Week 102
Population: The immunogenicity population for the core period included all participants who had received at least one dose of aducanumab in the core period and had at least one post-dose sample evaluated for immunogenicity in the core period. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aducanumab
Number analyzed (Participants) | 1595
Participants | 19

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to last follow-up visit (up to Week 170)
Description: The safety population included all participants who had received at least one dose of aducanumab in this study (221AD304).
Arm/Group | Aducanumab
All-Cause Mortality (participants affected / at risk) | 37/1696
Serious Adverse Events (participants affected / at risk) | 416/1696
Other Adverse Events (participants affected / at risk) | 1351/1696
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aducanumab (N=1696)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 13
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 5
Atrioventricular block second degree (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 7
Cardiac failure (Cardiac disorders) | 4
Cardiac failure chronic (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Pericarditis (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricle rupture (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 3
Retinal detachment (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 5
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Large intestine polyp (Gastrointestinal disorders) | 3
Leukoplakia oral (Gastrointestinal disorders) | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 3
Oesophageal motility disorder (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 4
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 2
Malaise (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 2
Anaphylactic shock (Immune system disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cat scratch disease (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 5
Clostridium difficile colitis (Infections and infestations) | 4
Covid-19 (Infections and infestations) | 16
Covid-19 pneumonia (Infections and infestations) | 8
Cystitis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 4
Diverticulitis intestinal perforated (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Klebsiella urinary tract infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Neuroborreliosis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 10
Pneumonia aspiration (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Subdural abscess (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Urinary tract infection pseudomonal (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 2
Accident (Injury, poisoning and procedural complications) | 3
Accidental overdose (Injury, poisoning and procedural complications) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 59
Femoral neck fracture (Injury, poisoning and procedural complications) | 14
Femur fracture (Injury, poisoning and procedural complications) | 6
Forearm fracture (Injury, poisoning and procedural complications) | 1
Foreign body in urogenital tract (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 7
Humerus fracture (Injury, poisoning and procedural complications) | 3
Incisional hernia (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3
Multiple fractures (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 3
Rib fracture (Injury, poisoning and procedural complications) | 4
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 7
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2
Tooth injury (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Wrong product administered (Injury, poisoning and procedural complications) | 1
Colonoscopy (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign nipple neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 3
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 9
Autonomic nervous system imbalance (Nervous system disorders) | 1
Bell's palsy (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Cerebellar haematoma (Nervous system disorders) | 1
Cerebellar stroke (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dementia alzheimer's type (Nervous system disorders) | 4
Dementia of the alzheimer's type, with delirium (Nervous system disorders) | 1
Dementia with lewy bodies (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Idiopathic generalised epilepsy (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 9
Loss of consciousness (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 2
Myelopathy (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 13
Small fibre neuropathy (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 23
Transient global amnesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 8
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 10
Behaviour disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 7
Neuropsychological symptoms (Psychiatric disorders) | 1
Psychiatric decompensation (Psychiatric disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 2
Tic (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
End stage renal disease (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Breast haematoma (Reproductive system and breast disorders) | 1
Breast swelling (Reproductive system and breast disorders) | 1
Colpocele (Reproductive system and breast disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Loss of personal independence in daily activities (Social circumstances) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Internal haemorrhage (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aducanumab (N=1696)
Constipation (Gastrointestinal disorders) | 87
Diarrhoea (Gastrointestinal disorders) | 130
Fatigue (General disorders) | 98
Covid-19 (Infections and infestations) | 427
Nasopharyngitis (Infections and infestations) | 107
Urinary tract infection (Infections and infestations) | 122
Contusion (Injury, poisoning and procedural complications) | 92
Fall (Injury, poisoning and procedural complications) | 355
Weight decreased (Investigations) | 91
Arthralgia (Musculoskeletal and connective tissue disorders) | 158
Back pain (Musculoskeletal and connective tissue disorders) | 140
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 443
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 424
Dizziness (Nervous system disorders) | 146
Headache (Nervous system disorders) | 246
Superficial siderosis of central nervous system (Nervous system disorders) | 232
Anxiety (Psychiatric disorders) | 104
Cough (Respiratory, thoracic and mediastinal disorders) | 103
Hypertension (Vascular disorders) | 130

LIMITATIONS AND CAVEATS:
The study was terminated prematurely based on the sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04241068/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04241068/SAP_001.pdf